CLINICAL TRIAL: NCT05549037
Title: Progression Survival Time According to Time-of-Day (ToD) of Administration of Immunochemotherapy for Advanced Non-small Cell Lung Cancer: A Phase III Randomized Control Trial
Brief Title: Effect of Time-of-Day (ToD) for Immunochemotherapy on PFS in NSCLC
Acronym: PACIFIC15
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Hunan Province Tumor Hospital (Other)
Responsible Party: Principal Investigator, Yongchang Zhang, Director, Head of Medical Oncology, Principal Investigator, Clinical Professor, Hunan Province Tumor Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: INJECTION
Record Dates: First submitted 2022-09-17; First posted 2022-09-22 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Non-small Cell Lung Cancer
Keywords: Immunochemotherapy; Time of day; Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — pembrolizumab; sintilimab

STUDY DESIGN:
Intervention Model Description: One for morning group, the patients in this group were treated with chemotherapy plus pembrolizumab or sintilimab before 15:00. One for afternoon group, the patients in this group were treated with chemotherapy plus pembrolizumab or sintilimab after 15:00.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A: Morning group (Experimental): All the patients in this arm will be treated with immunochemotherapy before 15:00.
  Interventions: Drug: Pembrolizumab, Sintilimab
- Arm B: Afternoon group (Experimental): All the patients in this arm will be treated with immunochemotherapy after 15:00.
  Interventions: Drug: Pembrolizumab, Sintilimab

INTERVENTIONS:
Drug: Pembrolizumab, Sintilimab — One for morning group, the patients in this group were treated with immunochemotherapy before 15:00. One for afternoon group, the patients in this group were treated with immunochemotherapy after 15:00.
  Other Names: time-of-day of administration of immunochemotherapy

SUMMARY:
This study aims to explore time-of-day of administration of immunochemotherapy on the efficacy for treatment naive advanced non-small cell lung cancer.

DETAILED DESCRIPTION:
All the advanced NSCLC patients who were treated with chemotherapy plus pembrolizumab or sitilimab will be randomized to two groups. One for morning group, the patients in this group were treated with chemotherapy plus pembrolizumab or sintilimab before 15:00. One for afternoon group, the patients in this group were treated with chemotherapy plus pembrolizumab or sintilimab after 15:00.

ELIGIBILITY:
Inclusion Criteria:

1. Understand the requirements and contents of the clinical trial, and provide a signed and dated informed consent form.
2. Age ≥ 18 years.
3. Histopathology or cytology confirmed and recorded local progression or metastatic non-small cell lung cancer without systemic treatment.
4. EGFR, ALK and ROS1 mutations negative confirmed by an accredited local laboratory.
5. ECOG 0-1.
6. Predicted survival ≥ 12 weeks.
7. Adequate bone marrow hematopoiesis and organ function
8. Presence of measurable lesions according to RECIST 1.1.
9. Subjects with stable brain metastases may be included in the study.

Exclusion Criteria:

1. Prior systemic therapy for locally advanced or metastatic disease.
2. Subjects who have received any of the following treatments must be excluded:

   * Ant Treatment with chemotherapy or molecules such as EGFR, VEGFR antibodies within 4 weeks prior to the first dose of study drug.
   * Have received radiation within 14 days prior to the first dose or have not recovered from radiation-related toxicity. Chest and extra-brain palliative radiotherapy, stereotactic radiosurgery, and stereotactic body radiotherapy may be performed 7 days prior to the first dose.
3. Presence of spinal cord compression or meningeal metastasis.
4. History of other malignant tumors within 2 years.
5. Adverse events (except alopecia of any degree) of CTCAE > grade 1 due to prior treatment (e.g., adjuvant chemotherapy, radiotherapy, etc.) prior to the first dose.
6. History of stroke or intracranial hemorrhage within 6 months prior to the first dose.
7. The presence of any severe or poorly controlled systemic disease, including poorly controlled hypertension and active bleeding in the judgment of the investigator.
8. Subjects with persistent or active infection, including but not limited to hepatitis B (HBV), hepatitis C (HCV), human immunodeficiency virus (HIV) and COVID-19 infection.
9. Heart-related diseases or abnormalities
10. Past history of interstitial lung disease, drug-induced interstitial lung disease, radiation pneumonitis requiring steroid therapy or interstitial lung disease with active clinical symptoms, immune pneumonia caused by immunotherapy.
11. Refractory nausea and vomiting, chronic gastrointestinal disease, difficulty swallowing drugs, or inability to adequately absorb sunvozertinib or anlotinib due to previous bowel resection.
12. Live vaccine was given 2 weeks before the first medication.
13. Women who are breastfeeding or pregnant.
14. Hypersensitivity to the test drug and the ingredients.
15. Other conditions assessed by the investigator to be unsuitable for participation in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Estimated)
Dates: Start 2022-09-23 (Actual); Primary Completion 2024-12-02 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | Time from first subject dose to study completion, or up to 36 month.
  To assess progression-free survival of patients treated by immunochemotherapy according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 by investigator, define as first dose to first documented disease progression assessed by investigator or death due to any cause.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | Time from first dose to last dose, or up to 24 month.
  To assess immunochemotherapy overall response rate according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 by investigator, define as the proportion of subjects who have a complete response (CR) or a partial response (PR)
Overall survival (OS) | Time from first subject dose to study completion, or up to 24 month.
  To assess overall survival, define as first dose to the death of the subject due to any cause.
Duration of Response (DoR) | Time from first subject dose to study completion, or up to 24 month.
  To assess duration of response for subjects with CR or PR according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 by investigator , defined as the time from the first documented CR or PR to disease progression or death

CONTACTS AND LOCATIONS:
Overall Officials: Yongchang Zhang, MD, Principal Investigator — Hunan Cancer Hospital
Locations (1):
- Hunan Cancer Hospital, Changsha, Hunan, China

REFERENCES:
- [Derived] Huang Z, Zeng L, Ruan Z, Zeng Q, Yan H, Jiang W, Xiong Y, Zhou C, Yang H, Liu L, Dai J, Zou N, Xu S, Wang Y, Wang Z, Deng J, Chen X, Wang J, Xiang H, Li X, Duchemann B, Chen G, Xia Y, Mok T, Scheiermann C, Levi F, Yang N, Zhang Y. Time-of-day immunochemotherapy in nonsmall cell lung cancer: a randomized phase 3 trial. Nat Med. 2026 Feb 2. doi: 10.1038/s41591-025-04181-w. Online ahead of print. PMID 41629425